CLINICAL TRIAL: NCT04532918
Title: An Open-label, 3-Treatment, 3-Period, Fixed Sequence Study in Healthy Subjects to Assess the Pharmacokinetics of Verinurad and Allopurinol When Administered Alone, and in Combination With Single Doses of Cyclosporine or Rifampicin
Brief Title: Pharmacokinetics of Verinurad and Allopurinol in Combination With Cyclosporine and Rifampicin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D5495C00013
Record Dates: First submitted 2020-08-04; First posted 2020-08-31 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-06

CONDITIONS: Chronic Kidney Disease
Keywords: Pharmacokinetics; Cyclosporine; Rifampicin; Drug-Drug interaction; Organic anion transporting polypeptide (OATP1B) 1
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — verinurad; Allopurinol; Cyclosporine; Rifampin

STUDY DESIGN:
Intervention Model Description: Fixed-sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Verinurad + allopurinol (Experimental): The subjects will receive single oral dose of verinurad 7.5 mg and allopurinol 300 mg under fasted condition.
  Interventions: Drug: Verinurad; Drug: Allopurinol
- Verinurad + allopurinol + cyclosporine (Experimental): The subjects will receive single oral dose of verinurad 7.5 mg, allopurinol 300 mg and cyclosporine 600 mg under fasted condition.
  Interventions: Drug: Verinurad; Drug: Allopurinol; Drug: Cyclosporine
- Verinurad + allopurinol + rifampicin (Experimental): The subjects will receive single oral dose of verinurad 7.5 mg, allopurinol 300 mg and rifampicin 600 mg under fasted condition.
  Interventions: Drug: Verinurad; Drug: Allopurinol; Drug: Rifampicin

INTERVENTIONS:
Drug: Verinurad — The subjects will receive single oral dose of extended release capsule verinurad 7.5 mg on Day 1 of each treatment period under fasted condition.
Drug: Allopurinol — The subjects will receive single oral dose of tablet allopurinol 300 mg on Day 1 of each treatment period under fasted condition.
Drug: Cyclosporine — The subjects will receive single oral dose of soft capsule cyclosporine 600 mg on Day 1 of treatment period 2 under fasted condition.
  Other Names: Sandimmun Optoral
  Arms: Verinurad + allopurinol + cyclosporine
Drug: Rifampicin — The subjects will receive single oral dose of film coated tablets rifampicin 600 mg on Day 1 of treatment period 3 under fasted condition.
  Other Names: Eremfat
  Arms: Verinurad + allopurinol + rifampicin

SUMMARY:
This Phase 1 study aims to quantify the effects of cyclosporine, a broad transporter inhibitor, and rifampicin, an OATP1B1/3 inhibitor, on verinurad pharmacokinetics (PK). The study is conducted in accordance with Food and Drug Administration guidance on Clinical Drug Interaction Studies, 2020. Verinurad will be developed as a fixed combination since it will always be administered together with allopurinol.

DETAILED DESCRIPTION:
This Phase 1 study will be an open-label, 3-period, 3-treatment, fixed-sequence study in healthy subjects (males and females of non-childbearing potential), performed at a single Clinical Unit.

The study will comprise of the following periods (visits):

* A Screening Period (Visit 1);
* A fixed sequence of 3 Treatment Periods during which subjects will be resident at the Clinical Unit from one day prior to administration of verinurad+allopurinol (Day -1) of Treatment Period 1 until the morning of Day 5 of the Treatment Period 2, and similarly for Treatment Period 3. There will be a washout period between Treatment Periods 2 and 3 dosing. The 3 Treatment Periods, include the washout period (Visits 2 to 3);
* A Follow-up Visit, after the last administration of verinurad+allopurinol (Visit 4).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent form prior to any study specific procedures.
* Healthy male or female subjects aged 18 - 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* Females must be either (1) Of non-childbearing potential, confirmed at Screening by fulfilling one of the following criteria (i) Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and Follicle-stimulating hormone (FSH) levels in the post-menopausal range (FSH >40 IU/mL).

(ii) Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

* Male subjects must adhere to the contraception methods.
* Have a body mass index between 18 and 30 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive).
* Must be able to swallow multiple capsules/tablets.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* Subject has a positive test result for severe acute respiratory syndrome coronavirus 2 before dosing in Treatment Period 1.
* Has clinical signs and symptoms consistent with coronavirus disease 2019 (COVID-19) infection, eg fever, dry cough, dyspnea, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* History of severe COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated).
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks prior to the first administration of verinurad.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at Screening (Visit 1) and on first admission (Day -1 in Treatment Period 1) as judged by the Investigator, including:

Alanine aminotransferase >1.5 × Upper limit of normal (ULN) Aspartate aminotransferase >1.5 × ULN Bilirubin (total) >1.5 × ULN Gamma glutamyl transpeptidase >1.5 × ULN If any of these tests are out of range, the test can be repeated once at the Screening Visit at the discretion of the Investigator.

* Any clinically significant abnormal findings in vital signs at Screening Visit and/or on admission (Day -1 in Treatment Period 1) to the Clinical Unit, including, but not limited to, any of the following:

  1. Systolic blood pressure <90 mmHg or >140 mmHg and/or diastolic blood pressure <50 mmHg or >90 mmHg sustained for more than 10 minutes while resting in a supine position
  2. Heart rate (resting, supine) <50 or >90 bpm
* Any clinically significant abnormalities on 12-lead electrocardiogram at Screening Visit, as judged by the Investigator, including, but not limited to any of the following:

  1. QTcF > 450 ms or < 340 ms or family history of long QT syndrome,
  2. Any significant arrhythmia,
  3. Conduction abnormalities,
  4. Clinically significant PR(PQ) interval prolongation (> 240 ms); intermittent second or third degree atrioventricular (AV) block, or AV dissociation,
  5. Complete bundle branch block and/or QRS duration > 120 ms.
* Any positive result at Screening Visit for serum hepatitis B surface antigen or anti-hepatitis B core antibody, hepatitis C antibody, and human immunodeficiency virus antibody.
* Suspicion or known Gilbert's and/or Lesch-Nyhan syndrome
* History of hypersensitivity to drugs with a similar chemical structure or class to verinurad, allopurinol, cyclosporine or rifampicin or excipients.
* Subjects who wear soft contact lenses (due to possible staining from rifampicin), unless the subject is prepared to refrain from wearing soft lenses throughout Treatment Period 3 until after the last PK sample collection.
* Women of childbearing potential.
* Carrier of the Human leukocyte antigen B*58:01 allele.
* Has received another new chemical or biological entity (defined as a compound which has not been approved for marketing in the US or EU) within 30 days or within 5 half-lives (whichever is longer) of the first administration of verinurad in this study.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to Novel uric acid transporter 1 transporter inhibitor & xanthine oxidase inhibitor.
* Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
* Positive screen for drugs of abuse, cotinine or alcohol at Screening or on each admission to the Clinical Unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of verinurad.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the Investigator. Excessive intake of alcohol defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g of alcohol per day for women.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the Investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day or would likely be unable to refrain from the use of caffeine-containing beverages during in-house stay at the investigational site.
* Involvement of any AstraZeneca, Parexel or Clinical Unit employee or their close relatives.
* Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who are vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the Investigator and/or are not able to read, speak and understand the German language.
* Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kӧrnicke, MD, Principal Investigator — Parexel Early Phase Clinical Unit Berlin
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP and SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00013&attachmentIdentifier=902e99d7-4601-4bca-8fd0-81e78c6be4ba&fileName=D5495C00013_CSP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 10-Sep-2020 and 23-Nov-2020 in Germany.
Pre-assignment Details: Participants who met the inclusion and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- Overall Study: Participants received treatments in 3 different treatment periods. Single oral dose of extended release capsule verinurad 7.5 mg, and tablet allopurinol 300 mg, in all 3 treatment periods, under fasted conditions. Along with, participants also received single oral dose of soft capsule of cyclosporine 600 mg in treatment period 2, and film coated tablets of rifampicin 600 mg in treatment period 3 respectively, under fasted condition. There was a washout period of 14 days between treatment periods 2 and 3 dosing.
Period: Overall Study
Arm/Group | Overall Study
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug, and for whom safety post-dose data were available, were included in the safety analysis for the study.
Arm/Group | Overall Study
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratio of Maximum Observed Plasma Peak Concentration (Cmax) for Verinurad
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of verinurad. Verinurad Cmax ratio of geometric mean of test treatment (verinurad+allopurinol with [cyclosporine or rifampicin], relative to reference treatment (verinurad+allopurinol alone) in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: The pharmacokinetic (PK) analysis set included all participants in the safety analysis set who received a verinurad+allopurinol dose and who had at least 1 quantifiable post-dose plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Period 1: Verinurad + Allopurinol: Participants received a single oral dose extended release capsule of verinurad 7.5 mg, and tablet of allopurinol 300 mg, under fasted conditions from days 1 to 5.
- Period 2: Verinurad + Allopurinol + Cyclosporine: Participants received a single oral dose extended release capsule verinurad 7.5 mg, tablet allopurinol 300 mg, and soft capsule cyclosporine 600 mg, under fasted conditions from days 1 to 5.
- Period 3: Verinurad + Allopurinol + Rifampicin: Participants received a single oral dose extended release capsule verinurad 7.5 mg, tablet allopurinol 300 mg, and film coated tablets rifampicin, under fasted conditions from days 1 to 5.
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
ng/mL | 13.30 (53.48) | 33.96 (29.39) | 26.09 (32.28)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of Cmax; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 255.3, 90% CI 2-sided [208.7 to 312.3] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of Cmax; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 189.5, 90% CI 2-sided [154.0 to 233.1] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

2. Primary Outcome: Geometric Mean Ratio of Area Under Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) for Verinurad
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of verinurad. Verinurad AUCinf ratio of geometric means of test treatment, relative to reference treatment in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: The PK analysis set included all participants in the safety analysis set who received a verinurad+allopurinol dose and who had at least 1 quantifiable post-dose plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
h*ng/mL | 90.25 (50.76) | 215.1 (30.94) | 138.0 (26.11)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUCinf; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 238.4, 90% CI 2-sided [207.6 to 273.8] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of AUCinf; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 148.9, 90% CI 2-sided [129.1 to 171.7] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

3. Primary Outcome: Geometric Mean Ratio of Area Under the Plasma Concentration-time Curve From Zero to Time of Last Quantifiable Concentration (AUClast) for Verinurad
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of verinurad. Verinurad AUClast ratio of geometric means of test treatment, relative to reference treatment in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
h*ng/mL | 79.67 (50.43) | 208.6 (30.07) | 133.4 (26.59)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUClast; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 261.8, 90% CI 2-sided [229.8 to 298.1] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of AUClast; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 163.2, 90% CI 2-sided [142.8 to 186.6] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

4. Secondary Outcome: Geometric Mean Ratio of Cmax for Verinurad Metabolites: M1 and M8
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of verinurad metabolites M1 and M8. Cmax ratio of geometric means of test treatment, relative to reference treatment in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
ng/mL
  M1 | 17.24 (50.28) | 47.14 (34.05) | 48.70 (31.47)
  M8 | 15.57 (40.02) | 3.839 (59.94) | 6.002 (48.53)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of Cmax for metabolite: M1; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 273.4, 90% CI 2-sided [227.9 to 328.1] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of Cmax for metabolite: M1; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 275.9, 90% CI 2-sided [228.7 to 332.7] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)
Statistical Analysis 3: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of Cmax for metabolite: M8; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 24.65, 90% CI 2-sided [19.15 to 31.72] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 4: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of Cmax for metabolite: M8; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 37.82, 90% CI 2-sided [29.18 to 49.03] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

5. Secondary Outcome: Geometric Mean Ratio of AUCinf for Verinurad Metabolites: M1 and M8
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of verinurad metabolites M1 and M8. AUCinf ratio of geometric means of test treatment, relative to reference treatment in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
h*ng/mL
  M1 | 119.5 (50.57) | 348.7 (39.87) | 264.9 (30.04)
  M8 | 110.3 (46.28) | 60.98 (60.46) | 77.35 (43.24)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUCinf for metabolite: M1; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 291.8, 90% CI 2-sided [260.6 to 326.8] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of Cmax for metabolite: M1; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 215.8, 90% CI 2-sided [192.0 to 242.4] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)
Statistical Analysis 3: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUCinf for metabolite: M8; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 55.31, 90% CI 2-sided [47.19 to 64.83] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 4: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of AUCinf for metabolite: M8; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 68.28, 90% CI 2-sided [57.99 to 80.39] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

6. Secondary Outcome: Geometric Mean Ratio of AUClast for Verinurad Metabolites: M1 and M8
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of verinurad metabolites M1 and M8. AUClast ratio of geometric means of test treatment, relative to reference treatment in each treatment period is reported.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
h*ng/mL
  M1 | 111.6 (51.84) | 341.9 (40.12) | 260.6 (30.70)
  M8 | 101.8 (45.17) | 51.95 (52.12) | 73.23 (44.42)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUClast for metabolite: M1; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 306.4, 90% CI 2-sided [273.3 to 343.6] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of AUClast for metabolite: M1; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 227.4, 90% CI 2-sided [202.1 to 255.8] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)
Statistical Analysis 3: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUClast for metabolite: M8; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 51.03, 90% CI 2-sided [43.80 to 59.45] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 4: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of AUClast for metabolite: M8; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 70.45, 90% CI 2-sided [60.21 to 82.44] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

7. Secondary Outcome: Geometric Mean Ratio of Cmax for Allopurinol and Oxypurinol
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of allopurinol and oxypurinol. Cmax ratio of geometric means of test geometric means of test treatment, relative to reference treatment in each treatment period is reported.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
ng/mL
  Allopurinol | 1947 (51.09) | 1457 (33.20) | 1597 (38.55)
  Oxypurinol | 6064 (18.15) | 5876 (18.24) | 6051 (20.41)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of Cmax for allopurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 74.84, 90% CI 2-sided [59.42 to 94.26] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of Cmax for allopurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 80.99, 90% CI 2-sided [63.88 to 102.7] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)
Statistical Analysis 3: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of Cmax for oxypurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 96.86, 90% CI 2-sided [92.11 to 101.8] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 4: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of Cmax for oxypurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 99.07, 90% CI 2-sided [94.36 to 104.0] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

8. Secondary Outcome: Geometric Mean Ratio of AUCinf for Allopurinol and Oxypurinol
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of allopurinol and oxypurinol. AUCinf ratio of geometric means of test geometric means of test treatment, relative to reference treatment in each treatment period is reported.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
h*ng/mL
  Allopurinol | 3982 (22.69) | 3914 (20.06) | 4163 (19.24)
  Oxypurinol | 196500 (28.48) | 181900 (24.23) | 195500 (24.85)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUCinf for allopurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 98.29, 90% CI 2-sided [91.26 to 105.9] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of AUCinf for allopurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 101.2, 90% CI 2-sided [93.72 to 109.2] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)
Statistical Analysis 3: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUCinf for oxypurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 99.16, 90% CI 2-sided [95.02 to 103.5] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 4: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of AUCinf for oxypurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 96.05, 90% CI 2-sided [92.15 to 100.1] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

9. Secondary Outcome: Geometric Mean Ratio of AUClast for Allopurinol and Oxypurinol
Description: Evaluation of a single dose of cyclosporine or rifampicin on the PK of allopurinol and oxypurinol. AUClast ratio of geometric means of test geometric means of test treatment, relative to reference treatment in each treatment period is reported.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
h*ng/mL
  Allopurinol | 3889 (23.01) | 3821 (19.78) | 4080 (19.24)
  Oxypurinol | 183600 (24.64) | 170600 (22.29) | 182100 (21.72)
Statistical Analysis 1: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUClast for allopurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 98.25, 90% CI 2-sided [91.10 to 106.0] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 2: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Statistical comparison of AUClast for allopurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 101.6, 90% CI 2-sided [93.99 to 109.8] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)
Statistical Analysis 3: Comparison: Period 1: Verinurad + Allopurinol vs Period 2: Verinurad + Allopurinol + Cyclosporine; Statistical comparison of AUClast for oxypurinol; Test type: Other — Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Geometric Mean Ratio (%) = 98.05, 90% CI 2-sided [94.50 to 101.7] — Pairwise comparisons of Test 1/ reference (verinurad+allopurinol+cyclosporine/ verinurad+allopurinol alone)
Statistical Analysis 4: Comparison: Period 1: Verinurad + Allopurinol vs Period 3: Verinurad + Allopurinol + Rifampicin; Analysis of variance of log transformed PK parameter with treatment and participant as fixed effects; Test type: Other; Geometric Mean Ratio (%) = 95.98, 90% CI 2-sided [92.61 to 99.48] — Pairwise comparisons of Test 2/ reference (verinurad+allopurinol+rifampicin/ verinurad+allopurinol alone)

10. Secondary Outcome: Area Under Plasma Concentration-time Curve From Zero to 24 Hours Post-dose AUC(0-24) of Verinurad, M1, M8, Allopurinol and Oxypurinol
Description: AUC(0-24) of verinurad, M1, M8, allopurinol and oxypurinol when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
h*ng/mL
  Verinurad | 62.02 (45.44) | 192.2 (31.45) | 118.4 (23.88)
  M1 | 86.23 (45.69) | 314.4 (39.75) | 242.9 (29.33)
  M8 | 79.80 (41.26) | 38.02 (45.54) | 48.81 (45.08)
  Allopurinol | 3982 (22.69) | 3914 (20.05) | 4163 (19.24)
  Oxypurinol | 100700 (17.92) | 95080 (18.15) | 98460 (18.59)

11. Secondary Outcome: Time to Reach Peak or Maximum Plasma Concentration (Tmax) for Verinurad, M1, M8, Allopurinol and Oxypurinol
Description: tmax of verinurad, M1, M8, allopurinol and oxypurinol when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Hours
  Verinurad | 4.03 [3.00 to 8.00] | 5.00 [2.98 to 6.02] | 4.00 [3.00 to 6.00]
  M1 | 4.02 [3.00 to 10.00] | 5.98 [4.02 to 10.03] | 4.00 [4.00 to 6.02]
  M8 | 4.52 [4.00 to 8.00] | 8.00 [5.00 to 12.00] | 5.00 [4.00 to 7.98]
  Allopurinol | 0.50 [0.50 to 2.02] | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 3.00]
  Oxypurinol | 4.00 [0.50 to 6.03] | 4.00 [0.50 to 5.00] | 3.00 [0.50 to 5.02]

12. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration Time Curve (t½λz) of Verinurad, M1, M8, Allopurinol and Oxypurinol
Description: t½λz of verinurad, M1, M8, allopurinol and oxypurinol when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Hours
  Verinurad | 20.31 (12.02) | 14.73 (13.00) | 15.03 (12.54)
  M1 | 18.04 (10.81) | 13.05 (9.455) | 12.52 (7.010)
  M8 | 18.25 (8.326) | 21.90 (24.13) | 14.89 (6.948)
  Allopurinol | 1.210 (0.1427) | 1.261 (0.2790) | 1.170 (0.1052)
  Oxypurinol | 23.19 (6.361) | 22.36 (4.977) | 23.76 (5.641)

13. Secondary Outcome: Terminal Elimination Rate Constant (λz) of Verinurad, M1, M8, Allopurinol and Oxypurinol
Description: λz of verinurad, M1, M8, allopurinol and oxypurinol when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/Hours
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
1/Hours
  Verinurad | 0.03842 (49.71) | 0.06101 (82.31) | 0.05557 (62.04)
  M1 | 0.04293 (47.35) | 0.06518 (71.96) | 0.06417 (61.89)
  M8 | 0.04163 (46.83) | 0.04497 (93.89) | 0.05133 (48.74)
  Allopurinol | 0.5770 (12.51) | 0.5616 (21.69) | 0.5950 (9.540)
  Oxypurinol | 0.03086 (26.32) | 0.03169 (22.14) | 0.02990 (23.34)

14. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma After Extravascular Administration (CL/F) for Verinurad and Allopurinol
Description: CL/F for verinurad and allopurinol when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/Hours
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Liter/Hours
  Verinurad | 92.30 (43.40) | 36.32 (10.44) | 55.99 (14.00)
  Allopurinol | 77.12 (17.51) | 78.09 (16.07) | 73.29 (14.24)

15. Secondary Outcome: Mean Residence Time of the Unchanged Drug in the Systemic Circulation (MRTinf) for Verinurad and Allopurinol
Description: MRTinf for verinurad and allopurinol when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Hours
  Verinurad | 21.28 (49.56) | 11.05 (50.07) | 12.60 (36.82)
  Allopurinol | 2.316 (30.10) | 2.713 (22.05) | 2.496 (20.04)

16. Secondary Outcome: Volume of Distribution (Apparent) at Steady State Following Extravascular Administration (Vss/F) of Verinurad and Allopurinol
Description: Vss/F of verinurad and allopurinol when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Liters
  Verinurad | 1768 (53.52) | 385.2 (52.45) | 685.0 (38.16)
  Allopurinol | 174.5 (41.88) | 208.0 (17.39) | 179.9 (30.55)

17. Secondary Outcome: Volume of Distribution (Apparent) at Steady State Following Extravascular Administration (Based on the Terminal Phase) (Vz/F) of Verinurad and Allopurinol
Description: Vz/F of verinurad and allopurinol when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Liters
  Verinurad | 2455 (1337) | 721.8 (574.6) | 1153 (758.7)
  Allopurinol | 133.5 (27.94) | 137.9 (20.16) | 122.6 (18.84)

18. Secondary Outcome: Metabolite:Parent (MP) Cmax Ratios for M1 and M8: Verinurad
Description: Metabolite:parent (MP) Cmax ratios for M1 and M8: verinurad when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Ratio
  M1: verinurad | 1.296 (36.79) | 1.388 (28.01) | 1.866 (24.09)
  M8: verinurad | 1.171 (30.12) | 0.1130 (56.62) | 0.2300 (52.89)

19. Secondary Outcome: Metabolite:Parent (MP) AUCinf Ratios for M1 and M8: Verinurad
Description: Metabolite:parent (MP) AUCinf ratios for M1 and M8: verinurad when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Ratio
  M1:verinurad | 1.324 (35.14) | 1.621 (23.80) | 1.919 (22.89)
  M8:verinurad | 1.222 (27.85) | 0.2834 (56.73) | 0.5604 (36.82)

20. Secondary Outcome: Metabolite:Parent (MP) AUClast Ratios for M1 and M8: Verinurad
Description: Metabolite:parent (MP) AUClast ratios for M1 and M8: verinurad when verinurad+allopurinol administered alone or in combination with cyclosporine or rifampicin in each treatment period.
Time Frame: Days 1 to 5 (pre-dose and post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Ratio
  M1:verinurad | 1.400 (28.68) | 1.639 (24.98) | 1.955 (23.27)
  M8:verinurad | 1.278 (26.07) | 0.2491 (54.22) | 0.5491 (39.93)

21. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: Assessment the safety and tolerability of verinurad and allopurinol in combination with cyclosporine or rifampicin
Time Frame: From screening (Day -28 to -2) until Follow-up or Early Termination (7-14 days after last verinurad dose)
Population: The safety analysis set included all participants who received at least 1 dose of study drug, and for whom safety post-dose data were available, were included in the safety analysis for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
Number analyzed (Participants) | 14 | 14 | 13
Participants
  Any AE | 2 | 10 | 3
  Any AE with outcome = death | 0 | 0 | 0
  Any SAE | 0 | 0 | 1
  Any AE leading to discontinuation of study drug | 0 | 1 | 0
  Any AE leading to withdrawal from study | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From screening (Day -28 to -2) until Follow-up or Early Termination (7-14 days after last verinurad dose)
Arm/Group | Period 1: Verinurad + Allopurinol | Period 2: Verinurad + Allopurinol + Cyclosporine | Period 3: Verinurad + Allopurinol + Rifampicin
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 1/13
Other Adverse Events (participants affected / at risk) | 2/14 | 10/14 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Verinurad + Allopurinol (N=14) | Period 2: Verinurad + Allopurinol + Cyclosporine (N=14) | Period 3: Verinurad + Allopurinol + Rifampicin (N=13)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Verinurad + Allopurinol (N=14) | Period 2: Verinurad + Allopurinol + Cyclosporine (N=14) | Period 3: Verinurad + Allopurinol + Rifampicin (N=13)
Feeling hot (General disorders) | 0 (0) | 8 (8) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT04532918/Prot_SAP_000.pdf